CLINICAL TRIAL: NCT04566458
Title: Real-World Data Study in HER2+ Metastatic Breast Cancer Patients in Third-Line Therapy
Brief Title: RWD Study in HER2+ mBC Patients in Third-Line Therapy
Status: Completed | Type: Observational
Sponsor: Exactis Innovation (Other)
Collaborators: Knight Therapeutics (Unknown)
Responsible Party: Sponsor
Other Study IDs: Exactis-05
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer Stage IV
Keywords: HER2 positive; Real World Data; Metastatic Breast cancer; Real World Evidence
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single arm: Her2 positive mBC patients who have received at least 3 lines of treatment in the metastatic setting.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — retrospective chart review study
  Other Names: No treatment was administered

SUMMARY:
This retrospective observational study will collect Canadian real-world data (RWD) from HER2+ metastatic breast cancer (mBC) patients to describe treatment sequences of all therapies received in the metastatic setting, to measure overall survival (OS), progression free survival (PFS), time to next active anti-cancer therapy, and to estimate the health resources utilization (HRU) during third-line therapy.

DETAILED DESCRIPTION:
The proportion of treatment received during all lines of therapy in the metastatic setting will be described. The 2-year survival rate and median OS with interquartile range (IQR) for third-line therapy will be calculated. HRU data and costs during third-line therapy will be collected.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients (≥18 years of age)

Patients with stage IV breast cancer

Patients with HER2+ status in metastatic setting

Patients that received at least two lines of active anti-cancer drugs due to disease progression.

Patients that began third-line therapy prior to October 31, 2018.

Exclusion Criteria:

Patients treated with an investigational anticancer agent in the ≥ 3rd line setting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population in this study will include up to 100 patients with HER2+ mBC having completed at least two previous lines of anti-HER2 based therapy or a combination of anti-HER2 based therapy and chemotherapy and ongoing third or additional lines of treatment.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
To describe treatment sequences of all lines of therapy received by HER2 + mBC patients in Canada | up to 2 years
  The proportion of each type of treatment received for all lines of therapy in the metastatic setting will be determined.
To describe the brain metastatic HER2+ mBC subpopulation during third line | up to 2 years
  The proportion of HER2+ mBC having brain metastasis at start of third lineas well as number of patients developing brain metastasis during third line will be quantified.
To describe radiation therapies received for brain metastasis in HER2+ mBC during third line. | up to 2 years
  The proportion of each type of radiation therapy received during third line, the time between brain metastasis detection and whole brain radiation (WBR), and the proportion of patients receiving a second WBR before death will be quantified.
To calculate the median overall survival (OS) of HER2+ mBC patients who received third-line therapy in Canada. | up to 2 years
  The 2-year survival rate and median OS in third-line HER2+ mBC patients will be quantified.
To calculate the median PFS of HER2+ mBC patients receiving third-line therapy in Canada | up to 2 years
  The median PFS in third-line HER2+ mBC patients will be quantified.
To calculate the median time to next active anticancer treatment of HER2+ mBC patients receiving third-line therapy in Canada | up to 2 years
  The median time to next active anticancer treatment in third-line HER2+ mBC patients will be quantified .
To assess HRU for HER2+ mBC patients in Canada during third-line therapy. | up to 2 years
  Information regarding HRU from HER2+ mBC patients in Canada during third-line therapy will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Batist, Principal Investigator — Exactis Innovation
Locations (8):
- Canada (8):
  - Centre hospitalier universitaire Dr-Georges-L.-Dumont, Moncton, New Brunswick
  - The Moncton Hospital, Moncton, New Brunswick
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Center, Toronto, Ontario
  - CHUM- Centre hospitalier de l'universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - CHUQ- Centre hospitalier universitaire de Québec, Québec, Quebec
  - CHUS-CIUSSS de l'Estrie - CHUS - Hôtel-Dieu and CHUS - Hôpital Fleurimont, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: Yes
The results of this retrospective observational study will not be formally documented in a Clinical Study Report. Coded patient-level data will be shared with the sponsor.